CLINICAL TRIAL: NCT05208112
Title: A Phase I Trial Evaluating the Safety, Tolerability and Pharmacokinetics of Intravenously Administered M6229 in Critically Ill Sepsis Patients - "HistoSeps"
Brief Title: Intravenously Administered M6229 in Critically Ill Sepsis Patients
Acronym: HistoSeps
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: A.P.J. Vlaar (Other)
Collaborators: Matisse Pharmaceuticals (Industry); Maastricht University (Other); Maastricht University Medical Center (Other)
Responsible Party: Sponsor-Investigator, A.P.J. Vlaar, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL77116.000.21
Record Dates: First submitted 2021-09-30; First posted 2022-01-26 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Sepsis; Septic Shock; Critical Illness
Keywords: sepsis; septic shock; histones; heparin; UFH; M6229; inflammation
MeSH Terms: conditions — Sepsis; Shock, Septic; Critical Illness; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: M6229 — Continuous intravenous infusion of M6229, a low-anticoagulant fraction of heparin. Dose-escalation is based on a modified continual reassessment method (mCRM) including escalation with overdose control (EWOC).

SUMMARY:
Sepsis is a life-threatening organ dysfunction caused by a dysregulated host response to infection. Mortality is high and survivors frequently suffer from long-term sequelae. Extracellular histones have been identified as essential mediators in the pathogenesis of sepsis and septic shock. These toxic molecules are released by damaged cells in response to infection and high extracellular levels can induce tissue injury and multiple organ dysfunction syndrome. Extracellular histones can be neutralized by complexation with the new candidate drug called M6229, a non-anticoagulant heparin, allowing the use of elevated dose levels relative to regular unfractionated heparin. This project aims at the roll-out of a first-in-man clinical study in sepsis patients evaluating the safety, tolerability, pharmacokinetics and pharmacodynamic effects of intravenously administered M6229 in subjects suffering from sepsis.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged ≥ 18 years old.
2. Signed informed consent by patient or legal representative.
3. Diagnosed with sepsis, defined by the Sepsis-3 criteria as a life-threatening organ dysfunction caused by a dysregulated host response to an infection.

   Organ dysfunction is defined by 1 of the following:

   a. Increase in SOFA score of ≥2. i. The baseline SOFA score can be assumed to be zero in patients not known to have pre-existing organ dysfunction.

   b. Acute kidney injury i. Defined as eGFR < 15 mL/min. c. Acute respiratory distress syndrome i. Defined by the Berlin criteria. d. The need of mechanical ventilation. e. Alteration in mental status.
4. The patients have to be included in the study within 72 hours of ICU admission due to sepsis or within 72 hours after sepsis diagnosis on the ICU. M6229 has to be administered within 84 hours after ICU admission due to sepsis or within 84 hours after sepsis diagnosis on the ICU.

Exclusion Criteria:

1. Subject has an advance directive to withhold life-sustaining treatments.
2. Subject is breastfeeding or intents to get pregnant within 30 days of enrolling into the study.
3. Subject is of childbearing potential and has a positive pregnancy test.

   a. A woman is considered to be of childbearing potential under the age of 60 years, unless surgically sterile.
4. Clinical suspicion or confirmation of a viral hemorrhagic shock syndrome including, but not limited to, dengue fever.
5. Bleeding risk:

   a. Clinical: i. Active bleeding; ii. Head trauma; iii. Intracranial surgery or stroke in the past 3 months; iv. History of intracerebral arteriovenous malformation, cerebral aneurysm or mass lesions of the central nervous system; v. Cerebral haemorrhage; vi. History of a bleeding diatheses; vii. Gastrointestinal bleeding in the past 6 weeks; viii. Presence of an epidural or spinal catheter; ix. Contraindication for IV therapeutic UFH. b. Laboratory: i. Platelet count <50 x109/L; ii. INR >2.0; iii. Baseline aPTT ≥45 seconds prior to enrolment, 1.5x upper limit of normal (ULN).
6. Use of any of the following treatments:

   1. UFH to treat a thrombotic event within 12 hours before infusion;
   2. LMWH within 24 hours before infusion;
   3. Warfarin (if used within 7 days before study entry AND if the INR exceeds 2.0 at enrolment);
   4. Direct oral anticoagulant (DOAC) use 3 days prior to enrollment.
   5. Thrombolytic therapy within 3 previous days;
   6. Use of IIb/IIIa inhibitors within the previous 7 days.
7. Confirmed antiphospholipid syndrome.
8. Known allergy to fish.
9. Cardiopulmonary resuscitation in the previous 7 days.
10. Liver failure defined as Child-Pugh Score Class C.
11. Abnormal liver function (ASAT and/or ALAT > 5 times upper limit of normal (ULN)).
12. Extracorporeal membrane oxygenation (ECMO) support dependent.
13. Pulmonary embolism or clinical suspicion of deep venous thrombosis (DVT).
14. Life expectancy of less than 24 hours.
15. Treating physician refusal.
16. Known adverse reaction to UFH, including heparin induced thrombocytopenia (HIT).
17. Participation in any other investigational drug study or other interventional study with interfering endpoints.
18. Any other clinical condition which, in the opinion of the investigator, would not allow safe completion of the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-04-05 (Actual); Primary Completion 2023-09-28 (Actual); Study Completion 2023-09-28 (Actual)

PRIMARY OUTCOMES:
aPTT changes before, during and after infusion of M6229 [Safety and tolerability] | Up to 72 hours after start infusion
  Anti-coagulation effects of M6229 determined by a change in aPTT at different time points during and after infusion of M6229.
Peak plasma concentration (Cmax) [Pharmacokinetics] | Up to 72 hours after start infusion
  Peak plasma concentration of M6229 in plasma
Steady state concentration (Css) [Pharmacokinetics] | Up to 72 hours after start infusion
  Steady state concentration of M6229 in plasma
Time to peak concentration (Tmax) [Pharmacokinetics] | Up to 72 hours after start infusion
  Time to peak concentration of M6229 in plasma
Area under the plasma concentration versus time curve (AUC) [Pharmacokinetics] | Up to 72 hours after start infusion
  Area under the plasma concentration versus time curve of M6229
Clearance [Pharmacokinetics] | Up to 72 hours after start infusion
  Clearance of M6229
Terminal half-life (t1/2) [Pharmacokinetics] | Up to 72 hours after start infusion
  Terminal half-life is the time required for the plasma concentration of M6229 to fall by 50% during the terminal phase
Volume of distribution (Vd) [Pharmacokinetics] | Up to 72 hours after start infusion
  Volume of distribution of M6229
Histone plasma level changes before, during and after infusion of M6229 [Efficacy] | Up to 72 hours after start infusion
  Change in histone plasma levels before and at different time-points after M6229 administration

SECONDARY OUTCOMES:
Incidence of excessive anti-coagulation effects [Safety and tolerability] | Up to 72 hours after start infusion
  Excessive anti-coagulation effects are:
  1. Clinical evidence or suspicion of severe non-surgical bleeding, defined as the administration of ≥ 2 units of blood products in 24 hours from start of infusion;
  2. aPTT > 90 seconds.
Incidence of adverse reactions [Safety and tolerability] | Up to 72 hours after start infusion
  Adverse reactions that are considered definitely and probably related to M6229 as specified in the protocol.
Changes in ECG corrected QT interval (QTc) [Safety and tolerability] | Up to 24 hours after start infusion
  Changes in ECGs QTc that are considered definitely and probably related to M6229
Amount of M6229 excreted in urine [Pharmacokinetics] | Up to 24 hours after start infusion
  Urine pharmacokinetic parameters of M6229 (amount of M6229 excreted in urine)
Change in plasma levels of D-Dimer before, during and after M6229 administration [Efficacy] | Up to 72 hours after start infusion
  Change in plasma levels of biomarkers of inflammation, coagulation and fibrinolysis (e.g. D-dimer, IL-6, IL-8) before and at different time-points after M6229 administration.
Change in plasma levels of interleukins before, during and after M6229 administration [Efficacy] | Up to 72 hours after start infusion
  Change in plasma levels of biomarkers of inflammation, coagulation and fibrinolysis (e.g. D-dimer, IL-6, IL-8) before and at different time-points after M6229 administration.
Correlation of histone plasma levels and abovementioned biomarkers with M6229 plasma levels (PK/PD) [Efficacy] | Up to 72 hours after start infusion
  Besides histone plasma levels, the investigators will also measure other biomarkers of inflammation, coagulation and fibrinolysis (e.g. D-dimer, IL-6, IL-8).
Severity of organ dysfunction based on Sequential Organ Failure Assessment (SOFA) score [Efficacy] | 30 days
  SOFA scores will be reported. Moreover, the investigators will compare these data with historic controls. For this, data will be used from a subset of patients included in a previously conducted study conducted in two tertiary teaching hospitals in the Netherlands named "Molecular Diagnosis and Risk Stratification of Sepsis" (MARS) study. The MARS study was a prospective observational study performed between January 2011 and January 2014 in the ICUs of the Amsterdam UMC, location AMC and UMC Utrecht.
Time on mechanical ventilation [Efficacy] | 30 days
  Ventilator free-days and time on mechanical ventilation. Data will be compared with historic controls from the MARS cohort.
Time on renal replacement therapy [Efficacy] | 30 days
  Renal replacement therapy free-days and time on renal replacement therapy. Data will be compared with historic controls from the MARS cohort.
Time on vasopression therapy [Efficacy] | 30 days
  Vasopressor free-days and time on vasopressors. Data will be compared with historic controls from the MARS cohort.
Length of stay [Efficacy] | 30 days
  ICU and hospital length of stays. Data will be compared with historic controls from the MARS cohort.
Mortality rate [Efficacy] | 30 days
  ICU and hospital mortality. Data will be compared with historic controls from the MARS cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander P Vlaar, MD, PhD, MBA, Principal Investigator — Department of Intensive Care Medicine, Amsterdam UMC, location AMC
Locations (2):
- Netherlands (2):
  - Maastricht UMC+, Maastricht, Limburg
  - Amsterdam UMC, location AMC, Amsterdam, North Holland

IPD SHARING:
Plan to Share IPD: No